CLINICAL TRIAL: NCT05728086
Title: Art Therapy to Address Hospital Clinician Burnout and Psychosocial Distress: a Randomised Controlled Trial
Brief Title: Art Therapy to Address Hospital Clinician Burnout
Acronym: CHArt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 316097
Record Dates: First submitted 2023-02-01; First posted 2023-02-14 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Burnout; Anxiety; Stress; Depression
Keywords: Art therapy; psychosocial distress; hospital clinicians; burnout
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Waitlist randomized controlled trial (RCT) design comprising an intervention group and a waitlist-control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group art therapy (Experimental): Participants randomised to the intervention group receive the group art therapy intervention shortly after baseline assessment. Adherence to the intervention will be checked via an adherence questionnaire completed by therapist delivering the intervention after each session. In addition, 20% of sessions will be observed by an independent researcher for adherence checking.
  Interventions: Other: Group art therapy
- waitlist control group (No Intervention): Participants randomised to the waitlist control group will complete outcomes measures at baseline and at the end of a 6 week waiting period. They will then begin the intervention (1-2 weeks after the intervention group has finished).

INTERVENTIONS:
Other: Group art therapy — The intervention is a manualised programme of group art therapy based on a bio-psychosocial therapeutic model. The programme is made up of six 60 - 90-minute art therapy group sessions facilitated by an experienced HCPC (Health and Care Professions Council) registered Art Therapists trained in the intervention.
  Arms: Group art therapy

SUMMARY:
A structured group art therapy intervention, comprising six 60 - 90-minute weekly workshops.

DETAILED DESCRIPTION:
The CHArt group art therapy intervention builds on a 6-week art therapy group intervention piloted with Barts Health oncology and palliative care doctors (Tjasink, M. 2019). It incorporates elements of workshops delivered for staff support by Barts art therapists during the Covid-19 pandemic (Tjasink, M., Stevens, P. 2022).

The intervention is broadly informed by affective neuroscience and evolutionary psychology theories with an emphasis on compassion-focused and resource-oriented therapeutic practice. Whilst the intervention draws on diverse influences, it aligns with the principles of Compassion Focussed Therapy (CFT), an integrative, bio-physiological psychological model underpinned by evolutionary theory.

Intervention elements include psycho-education, individual art making, collaborative group art making, art making in pairs, exploring a range of art materials and techniques (including clay, paint, natural objects and non-traditional mark - making materials), art-based grounding exercises and reflective discussion.

The intervention manual was developed by the study's Chief Investigator with input from a group of three art therapy experts (Health and Care Professions Council (HCPC) accredited art therapists working in National Health Service (NHS) medical contexts with experience of delivering art therapy - based staff support) and three experts by experience (Health Care professionals with experience of participating in art therapy - based staff support groups at work). Adherence to the intervention will be monitored through two adherence tools (therapist self reported and independent observer).

ELIGIBILITY:
Inclusion Criteria:

* • Healthcare professional employed in a patient facing clinical role by Barts Health NHS Trust or Barts Bank partners

  * 18 years or older
  * Willing and able to provide informed consent
  * Able to attend the group intervention sessions
  * Moderate to severe risk scored on any of the three MBI - HSS subscales or on the PSS 10:
  * emotional exhaustion score of ≥17, or
  * depersonalization score of ≥7, or
  * personal accomplishment score of ≤ 38 or
  * perceived stress (≥ 14)

Exclusion Criteria:

* • Unwilling or unable to give consent

  * Diagnosed with or treated for a serious depressive condition, a personality disorder or psychosis in the past 12 months. (Self-reporting through screening.)
  * Attempted suicide or made plans to commit suicide in the past 12 months. (Self-reporting through screening.)
  * Individual does not provide direct patient care for Barts Health NHS Trust

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Change in burnout element 'Emotional Exhaustion' assessed using the Emotional Exhaustion scale of The Maslach Burnout Inventory - Human Services Survey (MBI-HSS) | Baseline [T1], post 6-week intervention / post 6-week wait [T2], 12 week post intervention follow up [T3]
  The MBI-HSS assesses three elements of burnout syndrome: emotional exhaustion, depersonalization, and lack of personal accomplishment. Each element is measured by a separate scale. The Emotional Exhaustion (EE) scale assesses feelings of being emotionally over-extended and exhausted at work. It includes 9 items which are scored on a 7-item Likert scale from 0 = never to 6 = every day. The scale has a score range of 0-54 with higher scores corresponding to greater experiences of burnout.

SECONDARY OUTCOMES:
Change in burnout element 'depersonalisation' assessed using the Depersonalisation scale of The Maslach Burnout Inventory - Human Services Survey (MBI-HSS) | Baseline [T1], post 6-week intervention / post 6-week wait [T2], 12 week post intervention follow up [T3]
  Depersonalisation scale of the MBI - HSS
  The 5-item Depersonalization (DP) scale assesses an emotionally distant / indifferent response toward patients. It includes 6 items which are scored on a 7-item Likert scale from 0 = never to 6 = every day. The scale has a score range of 0-30 with higher scores corresponding to greater experiences of burnout.
Change in burnout element 'personal accomplishment' assessed using the Personal Accomplishment scale of The Maslach Burnout Inventory - Human Services Survey (MBI-HSS) | Baseline [T1], post 6-week intervention / post 6-week wait [T2], 12 week post intervention follow up [T3]
  Personal Accomplishment (PA) scale assesses feelings of competence and achievement in work with people. It includes 8 items which are scored on a 7-item Likert scale from 0 = never to 6 = every day. The scale has a score range of 0-48 with lower scores corresponding to greater experiences of burnout.
Change in anxiety assessed using the Generalised Anxiety Disorder Questionnaire (GAD 7) | Baseline [T1], post 6-week intervention / post 6-week wait [T2], 12 week post intervention follow up [T3]
  The GAD 7 assesses anxiety. It includes 7 items which are scored on a 4-item Likert scale from 0 = not at all to 3 = nearly every day. The scale has a score range of 0-21 with higher scores corresponding to greater levels of anxiety.
Change in depression assessed using the Personal Health Questionnaire Depression Scale (PHQ 8) | Baseline [T1], post 6-week intervention / post 6-week wait [T2], 12 week post intervention follow up [T3]
  The PHQ 8 assesses severity of depression. It includes 8 items which are scored on a 4-item Likert scale from 0 = not at all to 3 = nearly every day. The scale has a score range of 0-24 with higher scores corresponding to greater severity of depression.
Change in perceived stress assessed using the Perceived Stress Scale (PSS-10) | Baseline [T1], post 6-week intervention / post 6-week wait [T2], 12 week post intervention follow up [T3]
  The PSS10 assesses perceived stress. It includes 10 items which are scored on a 5-item Likert scale from 0 = never to 4 = very often. The scale has a score range of 0-40 with higher scores corresponding to greater levels of perceived stress.
CHArt Feedback Questionnaire | post 6-week intervention [T2]
  This is a participant experience feedback questionnaire. It includes 8 items on themes of perceived helpfulness, perceived behavioural change and attribution of change, barriers and enablers to attendance. Questions include multiple choice and follow - up free text elements. For example
  Question 6:
  Were there any barriers / challenges to attending?
  Yes, definitely; Yes, some; Not really; Not at all
  If so, what were they and how did you address them?
  If not, what made attendance possible for you?

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Priebe, Study Chair — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tjasink, M., G. Soosaipillai (2019) Art therapy to reduce burnout in oncology and palliative care doctors: a pilot study.
- [Background] Tjasink, M, Stevens, P. (2022). The innovative use of art psychotherapy with NHS clinicians in Jury, H. and Coles, A., 'Art Psychotherapy and Innovation: New Territories, Techniques and Technologies'. Jessica Kingsley, London: 83 - 103.
- [Background] Maslach, C. et al. (2018). Maslach burnout inventory: manual. [Menlo Park, Calif.], Mind Garden.
- [Derived] Tjasink M, Carr CE, Bassett P, Soosaipillai G, Ougrin D, Priebe S. Art therapy to reduce burnout and mental distress in healthcare professionals in acute hospitals: a randomised controlled trial. BMJ Public Health. 2025 Aug 3;3(2):e002251. doi: 10.1136/bmjph-2024-002251. eCollection 2025. PMID 40761359

DOCUMENTS (1):
  • Informed Consent Form (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT05728086/ICF_001.pdf